CLINICAL TRIAL: NCT01201811
Title: A Phase 4, Open-Label, Single-Arm Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Subcutaneous Azacitidine in Adult Taiwanese Subjects With Higher-Risk Myelodysplastic Syndromes.
Brief Title: Study of Azacitidine in Adult Taiwanese Subjects With Higher-Risk Myelodysplastic Syndromes (MDS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZA-MDS-001
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Results first posted 2014-06-24 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; Taiwan; Azacitidine; Vidaza; Celgene; Pathologic Processes; Neoplasms; Bone Marrow Diseases; Hematologic Diseases; Antineoplastic Agents; Antimetabolites, Antineoplastic; Antimetabolites; Molecular Mechanisms of Pharmacological Action; Pharmacologic Actions; Therapeutic Uses; Enzyme inhibitors
MeSH Terms: conditions — Myelodysplastic Syndromes; Pathologic Processes; Neoplasms; Bone Marrow Diseases; Hematologic Diseases | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-Arm (Experimental): Azacitidine 75 mg/m^2/day Subcutaneous for 7 days Day every 28 days for up to 6 cycles
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Subjects will receive azacitidine 75 mg/m2/day SC for 7 days every 28 days for up to 6 cycles, unless they are discontinued from the treatment. In addition, subjects may receive best supportive care as needed, including antibiotics and transfusions, per Investigator discretion.

SUMMARY:
The primary purpose of this study is to determine the effectiveness and safety of azacitidine in the treatment of Taiwanese subjects with higher-risk Myelodysplastic Syndrome (MDS).

DETAILED DESCRIPTION:
The study has 3 phases which include the Screening Phase, the Treatment Phase, and the Post-Treatment Phase and outlined as follows:

Screening Phase:

Subjects will provide informed consent prior to undergoing any study-related procedures. Screening procedures are to take place within 28 days prior to the initiation of azacitidine treatment (Day 1, Cycle 1). Subject eligibility will be based on central pathology review. Bone marrow aspirate and bone marrow biopsy will be collected at screening and sent for morphological assessment by a central pathology reviewer prior to the subject receiving IP. The central pathology reviewer will document the MDS classification according to the FAB and WHO criteria (Appendix A and B, respectively).

A standard cytogenetic metaphase preparation will be prepared from the bone marrow aspirate and sent to the local or central laboratory (for sites without local analysis capability) for the cytogenetic analysis prior to receiving IP.

The IPSS score will be calculated using the central reviewer's pathology report for bone marrow blast percentage, local cytogenetic assessment for karyotype, and central laboratory report for number of cytopenias (Appendix D).

Treatment Phase:

The first dose of azacitidine for each subject begins on Day 1 of Cycle 1. All subjects will receive azacitidine 75 mg/m2/day SC for 7 days every 28 days for up to 6 cycles, unless they are discontinued from treatment. Visits during the treatment phase are to be scheduled weekly for the first 2 cycles, then every other week for all subsequent cycles throughout the rest of the study. Safety and efficacy measures are to be performed weekly, every other week, every 4 weeks, or at 24 weeks, depending on the procedure.

Post-Treatment Phase:

All discontinued subjects, regardless of reason for discontinuation, should undergo end-of-study procedures at the time of study discontinuation. Subjects will have a follow-up visit for the collection of adverse events up to 28 days after last IP dose.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of RAEB or RAEB-T according to FAB classification for MDS and with an IPSS score of intermediate-2 or high risk or a diagnosis of myelodysplastic CMML per modified FAB criteria.
* Taiwanese males and females ≥ 18 years of age
* ECOG 0, 1, or 2;
* Adequate hepatic and renal organ function

Exclusion Criteria:

* Previous treatment with azacitidine or decitabine
* Malignant disease diagnosed within prior 12 months
* Uncorrected red cell folate deficiency or vitamin B12 deficiency
* Diagnosis of metastatic disease
* Malignant hepatic tumors
* Known or suspected hypersensitivity to azacitidine or mannitol
* Prior transplantation or cytotoxic therapy, including azacitidine and chemotherapy, administered to treat MDS
* Treatment with erythropoietin or myeloid growth factors during the 21 days prior to Day 1 of Cycle 1 or androgenic hormones during the 14 days prior to Day 1 of Cycle 1;
* Active HIV or viral hepatitis type B or C
* Treatment with other investigational drugs within the previous 30 days prior to Day 1 of Cycle 1, or ongoing adverse events from previous treatment with investigational drugs, regardless of the time period;
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C L Beach, PharmD, Study Director — Celgene
Locations (11):
- Taiwan (11):
  - Changhua Christian Hospital, Changhua
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Buddhist Tzu Chi General Hospital-Hualien Tzu Chi Medical Center, Hualien City
  - Kaohsiung Medical Hospital University, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Shuang-ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei

REFERENCES:
- [Background] Chou WC, Yeh SP, Hsiao LT, Lin SF, Chen YC, Chen TY, Laille E, Galettis A, Dong Q, Songer S, Beach CL. Efficacy, safety, and pharmacokinetics of subcutaneous azacitidine in Taiwanese patients with higher-risk myelodysplastic syndromes. Asia Pac J Clin Oncol. 2017 Oct;13(5):e430-e439. doi: 10.1111/ajco.12659. Epub 2017 Jan 25. PMID 28124500

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at nine investigational sites within Taiwan. The purpose of the current study was to evaluate the efficacy, safety, and steady-state Pharmacokinetic (PK) profile of subcutaneous (SC) azacitidine given at a dose of 75 mg/m^2/day for 7 days in Taiwanese participants with higher-risk Myelodysplastic Syndrome (MDS).
Groups:
- Azacitidine: Azacitidine 75 mg/m^2/day subcutaneously (SC) for 7 days every 28 days for up to 6 cycles
Period: Overall Study
Arm/Group | Azacitidine
Started | 44
Completed | 25
Not Completed | 19
Not completed — Adverse Event | 6
Not completed — Disease progression | 3
Not completed — Withdrawal by Subject | 3
Not completed — Death | 4
Not completed — Treatment Failure | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population was defined as all enrolled participants.
Arm/Group | Azacitidine
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Taiwanese origin
  Participants
    Asian | 44
Myelodysplastic Syndrome (MDS) French-American-British (FAB) Classification [Count of Participants; unit: Participants] — FAB is a classification system for five (5) subtypes of myelodysplastic syndrome that are distinguished by the percentage of myeloblasts, presence or absence of ringed sideroblasts or a monocytosis. Classification was made by the Local Reviewer.
  Participants
    Refractory anemia with excess blasts (RAEB) | 35
    RAEB in transformation | 7
    Chronic myelomonocytic leukemia (Modified CMML) | 2
    Acute myelogenous leukemia (AML) | 0
World Health Organization (WHO) Classification [Count of Participants; unit: Participants] — The World Health Organization (WHO) classification recognizes eight subtypes of MDS that are distinguished by the percentage of myeloblasts, presence or absence of ringed sideroblasts (i.e., erythroid precursors with iron deposits surrounding the nucleus), presence of a monocytosis or a deletion 5q.
  Participants
    Refractory anemia with excess blasts (RAEB-1) | 15
    Refractory anemia with excess blasts (RAEB-2) | 23
    Acute myelogenous leukemia (AML) | 5
    Chronic myelomonocytic leukemia (CMML -1) | 1
    Chronic myelomonocytic leukemia (CMML-2) | 0
    Refractory anemia (RA) | 0
    RA with ringed sideroblasts (RARS) | 0
    Refractory Cytopenia Multilineage Dysplasia (RCMD) | 0
    Myelodysplastic Syndrome - Unclassified (MDS-U) | 0
International Prognostic Scoring System (IPSS) [Count of Participants; unit: Participants] — The international prognostic scoring system (IPSS) is a standard for risk assessment in primary myelodysplastic syndromes (MDS) that categorizes prognoses taking into account cytogenetics, cytopenias, blasts and blood counts. The IPSS prognostic subgroups consist of low-, intermediate-1-, intermediate-2-, and high-risk groups. The scale is 0-3.5 at 0.5 increments. Scores of 0=Low; 0.5-1.0=Int-1; 1.5-2.0=Int-2; 2.5-3.5=High risk which corresponds to poorer prognosis. The assessment was performed by the local investigator
  Participants
    Low risk (0) | 0
    Intermediate-1 (0.5 - 1.0) | 2
    Intermediate-2 (1.5 - 2.0) | 16
    High Risk (≥ 2.5) | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Hematologic Response Using International Working Group (IWG) Criteria for Myelodysplastic Syndrome (MDS) and Assessed by Investigator
Description: Hematologic Response according to the 2000 International Working Group (IWG) response criteria for MDS was based on the Investigators determination and defined as:
  * Complete Response (CR): repeat bone marrow (BM) shows <5% myeloblasts, and peripheral blood values lasting ≥ 2 months of hemoglobin (hgb) (>110 g/L), neutrophils (≥1.5x10^9/L), platelets (≥100x10^9/L), blasts (0%) and no dysplasia
  * Partial Response (PR): same as CR for peripheral blood: BM shows blasts decrease by ≥ 50% or a less advanced FAB classification from pretreatment
  * Stable disease (SD): failure to achieve a PR, no evidence of progression for at least 2 months.
  * Failure: death during treatment or disease progression
  * Relapse After CR or PR: return to pretreatment BM blast percent or decrement of ≥ 50% from remission/response levels in granulocytes or platelets; or reduction in hgb by ≥20 g/L or transfusion dependence
  * Disease Progression: change in blast levels
  * Disease Transformation to AML
Time Frame: Response assessed at end of cycle 6; through week 24; End of study
Population: The intention-to-treat (ITT) population was defined as all enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 44
percentage of participants
  Overall (CR+PR) | 0 [0.0 to 8.0]
  Overall (CR+PR+SD) | 63.6 [47.8 to 77.6]
  Complete Remission (CR) | 0.0 [0.0 to 8.0]
  Partial Remission (PR) | 0.0 [0.0 to 8.0]
  Stable Disease (SD) | 63.6 [47.8 to 77.6]
  Disease Progression (DP) | 2.3 [0.1 to 12.0]
  Transformation to AML | 4.5 [0.6 to 15.5]
  Failure | 4.5 [0.6 to 15.5]
  No Response Assessed | 25.0 [13.2 to 40.3]

2. Primary Outcome: Percentage of Participants Showing Hematologic Improvement Using International Working Group (IWG Criteria for Hematologic Improvement Cheson 2000) Criteria for Myelodysplastic Syndrome (MDS) and Assessed by Sponsor
Description: Hematologic improvements (HI) have 4 categories:
  1. Erythroid response (HI-E): Major >20g/L increase or transfusion independent. Minor- 10-20g/L increase or ≥50% decrease in transfusion requirements.
  2. Platelet response (HI-P): Major absolute increase of ≥30x10^9/L or platelet transfusion independence. Minor-≥50% increase.
  3. Neutrophil response (HI-N): Major 100% increase or an absolute increase of >0.5x10^9/L. Minor-≥100% increase and absolute increase of <0.5x10^9/L
  4. Progression or relapse after HI
  Overall hematological improvement (HI) was defined as any type (major or minor) of improvement of HI-E, HI-P, or HI-N. Criteria: Pretreatment=hemoglobin <100g/L or RBC transfusion-dependent, platelet count <100x10^9/L or platelet transfusion dependent, absolute neutrophil count <1.5x10^9/L. Sponsor's determination was derived using clinically relevant data.
  Denominator for progression/relapse after HI included participants who had achieved HI.
Time Frame: Response assessed at end of cycle 6; through week 24; End of study
Population: The intention-to-treat (ITT) population was defined as all enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 44
percentage of participants
  Any improvement | 50.0 [34.6 to 65.4]
  Hematologic Improvement-E (major) | 31.8 [18.6 to 47.6]
  Hematologic Improvement-E (minor) | 9.1 [2.5 to 21.7]
  Hematologic Improvement-P (major) | 37.8 [22.5 to 55.2]
  Hematologic Improvement-P (minor) | 0 [0 to 9.5]
  Hematologic Improvement-N (major) | 7.1 [0.9 to 23.5]
  Hematologic Improvement-N (minor) | 0 [0 to 12.3]
  Progression/relapse after HI | 27.3 [10.7 to 50.2]

3. Other Pre Specified Outcome: Participants' Red Blood Cell (RBC) Transfusion Status for Participants Who Were Transfusion Dependent at Baseline
Description: A participant was considered transfusion dependent at baseline if the participant had one or more Red Blood Cell transfusions during the 56 days prior to first dose. During the study, a participant was considered transfusion independent during the on-treatment period if the participant had no transfusions during any 56 consecutive days or more (e.g., Day 1 through 56, Day 2 through 57, etc). Otherwise, they were considered transfusion dependent.
  The total N=44, but 1 participant can only be dependent or independent at baseline for each type of transfusion (ie, total = 44: RBC dependent at BL=32, RBC independent at BL=12)
Time Frame: Baseline to Cycle 6; The on-treatment period was considered the period from the date of the first dose to the last treatment study visit
Population: The intent-to-treat (ITT) participants who were transfusion dependent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 32
percentage of participants
  Baseline Dependent: On-Treatment Independent | 37.5 (1.97) [21.1 to 56.3]
  Baseline Dependent; On-Treatment Dependent | 62.5 (2.47) [43.7 to 78.9]

4. Other Pre Specified Outcome: Participants' Red Blood Cell (RBC) Transfusion Status for Participants Who Were Transfusion Independent at Baseline
Description: A participant was considered RBC transfusion-independent at baseline if the participant had no RBC transfusions during the 56 days prior to first dose. During the study, a participant was considered transfusion independent during the on-treatment period if the participant had no RBC transfusions during any 56 consecutive days or more (eg, Days 1 through 56, Days 2 through 57, etc.). Otherwise, they were considered transfusion dependent.
  The total N=44, but 1 participant can only be dependent or independent at baseline for each type of transfusion (ie, total = 44: RBC dependent at BL=32, RBC independent at BL=12)
Time Frame: as for outcome 3
Population: The Intent to Treat (ITT) participants who were transfusion independent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
percentage of participants
  Baseline Independent; On-Treatment Independent | 75.0 [42.8 to 94.5]
  Baseline Independent; On-Treatment Dependent | 25.0 [5.5 to 57.2]

5. Secondary Outcome: Number of Red Blood Cell (RBC) Transfusions by Cycle
Description: The number of transfusions received 56 days prior to treatment and during study were standardized per 28 days and summarized by cycle for RBCs. The formula for standardizing per 28 days was: [(# of transfusions in the measurement period / length of the measurement period (days)) x 28], where the measurement period was either baseline or the relevant cycle length. For each participant the overall post-baseline average was calculated as the average of # of RBC transfusions per cycle.
Time Frame: Up to week 24;The on-treatment period was considered the period from the date of the first dose to the last treatment study visit.
Population: ITT Population- The intent-to-treat (ITT) population was defined as all enrolled participants.
Measure: Mean (Standard Deviation); unit: Transfusions
Arm/Group | Azacitidine
Number analyzed (Participants) | 44
Transfusions
  Baseline (N = 44) | 1.3 (1.97)
  Overall Post-Baseline Average (N = 44) | 2.4 (2.47)
  overall Change from Baseline ( N = 44) | 1.0 (2.59)
  Cycle 1 ( N = 44) | 2.5 (2.27)
  Cycle 2: number analyzed (Participants) | 41
  Cycle 2 | 2.3 (2.03)
  Cycle 3: number analyzed (Participants) | 38
  Cycle 3 | 2.2 (2.90)
  Cycle 4: number analyzed (Participants) | 30
  Cycle 4 | 1.5 (2.11)
  Cycle 5: number analyzed (Participants) | 27
  Cycle 5 | 1.4 (2.59)
  Cycle 6: number analyzed (Participants) | 26
  Cycle 6 | 1.9 (3.96)

6. Other Pre Specified Outcome: Participants' Platelet Transfusion Status for Participants Who Were Transfusion Dependent at Baseline
Description: A participant was considered platelet transfusion dependent at baseline if the participant had one or more platelet transfusions during the 56 days prior to first dose. During the study, a participant was considered platelet transfusion independent during the on-treatment period if the participant had no platelet transfusions during any 56 consecutive days or more (eg, Days 1 through 56, Days 2 through 57, etc.). Otherwise, they were considered platelet transfusion dependent.
  The total N=44, but 1 participant can only be dependent or independent at baseline for each type of transfusion (ie, total = 44: platelet dependent at BL=18, platelet independent at BL=26)
Time Frame: as for outcome 3
Population: The intent-to-treat (ITT) population who were transfusion dependent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 18
percentage of participants
  Baseline Dependent; On-Treatment Independent | 38.9 [17.3 to 64.3]
  Baseline Dependent; On-Treatment Dependent | 61.1 [35.7 to 82.7]

7. Other Pre Specified Outcome: Participants' Platelet Transfusion Status for Participants Who Were Transfusion Independent at Baseline
Description: A participant was considered platelet transfusion independent at baseline if the participant had no platelet transfusions during the 56 days prior to first dose. During the study, a participant was considered platelet transfusion independent during the on-treatment period if the participant had no platelet transfusions during any 56 consecutive days or more (eg, Days 1 through 56, Days 2 through 57, etc.). Otherwise, they were considered platelet transfusion dependent.
  The total N=44, but 1 participant can only be dependent or independent at baseline for each type of transfusion (ie, total = 44: platelet dependent at BL=18, platelet independent at BL=26)
Time Frame: as for outcome 3
Population: The intent-to-treat (ITT) participants who were transfusion independent
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Azacitidine
Number analyzed (Participants) | 26
percentage of particpants
  Baseline Independent: On-Treatment Independent | 76.9 [56.4 to 91.0]
  Baseline Independent; On-Treatment Dependent | 23.1 [9.0 to 43.6]

8. Secondary Outcome: Number of Platelet Transfusions by Cycle
Description: The number of transfusions received 56 days prior to treatment and during study was standardized per 28 days and summarized by cycle for platelets. The formula for standardizing per 28 days was: [(# of transfusions in the measurement period / length of the measurement period (days)) x 28], where the measurement period was either baseline or the relevant cycle length. For each participant the overall post-baseline average was calculated as the average of # of platelet transfusions per cycle.
Time Frame: Up to week 24; The on-treatment period was considered the period from the date of the first dose to the last treatment study visit.
Population: The intent-to-treat (ITT) population was defined as all enrolled participants.
Measure: Mean (Standard Deviation); unit: Transfusions
Arm/Group | Azacitidine
Number analyzed (Participants) | 44
Transfusions
  Baseline ( N = 44) | 0.9 (2.40)
  Overall Post-Baseline Average ( N= 44) | 2.7 (3.56)
  OverallChange from Baseline ( N = 44) | 1.8 (3.53)
  Cycle 1 ( N = 44) | 2.6 (3.38)
  Cycle 2: number analyzed (Participants) | 41
  Cycle 2 | 2.3 (3.28)
  Cycle 3: number analyzed (Participants) | 38
  Cycle 3 | 3.0 (4.85)
  Cycle 4: number analyzed (Participants) | 30
  Cycle 4 | 1.6 (2.89)
  Cycle 5: number analyzed (Participants) | 27
  Cycle 5 | 1.9 (3.61)
  Cycle 6: number analyzed (Participants) | 26
  Cycle 6 | 2.7 (6.01)

9. Secondary Outcome: Number of Infections (Post-baseline Average) Requiring Intravenous Antibiotics, Anti-fungals, or Antivirals Per 28 Days
Description: The on-treatment adverse event of infection requiring IV antibiotics, antifungals, or antivirals per 28 days/cycle. The overall post-baseline average is the average of number of infections requiring IV antibiotics or IV antiviral per 28 days/cycle. For each participant the overall post-baseline average was calculated as the average of # of infections requiring IV antibiotics or IV antiviral per 28 days per cycle.
Time Frame: as for outcome 8
Population: The intent-to-treat (ITT) population was defined as all enrolled participants.
Measure: Mean (Standard Deviation); unit: Infections per cycle
Arm/Group | Azacitidine
Number analyzed (Participants) | 44
Infections per cycle
  Baseline | 0.1 (0.51)
  Overall Post Baseline | 0.5 (0.79)
  Overall Change from Baseline | 0.4 (0.98)
  Cycle 1 | 0.5 (0.85)
  Cycle 2 | 0.4 (0.61)
  Cycle 3 | 0.4 (0.82)
  Cycle 4 | 0.1 (0.39)
  Cycle 5 | 0.1 (0.38)
  Cycle 6 | 0.2 (0.66)

10. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE that resulted in any of the following outcomes was defined as a serious adverse event (SAE):
  * Death;
  * Life-threatening event;
  * Any inpatient hospitalization or prolongation of existing hospitalization;
  * Persistent or significant disability or incapacity;
  * Congenital anomaly or birth defect;
  * Any other important medical event.
  The severity of an AE was evaluated by the investigator according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (Version 4.0) where Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Death. Treatment Emergent AEs (TEAE) were defined as AEs with an onset date on or after the first dose of study drug and within 28 days after the date of the last dose. In addition, any AE that occurred beyond this timeframe and that was assessed by the investigator as possibly related to study drug was considered a TEAE.
Time Frame: From the first dose of study drug through 28 days after completion of/discontinuation from the study (maximum time on study drug 244 days)
Population: Safety Population included enrolled participants who received at least one dose of investigational product and had at least one postdose assessment
Measure: Number; unit: participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 44
participants
  ≥ 1 TEAE | 44
  ≥ 1 NCI Grade 3 or 4 TEAE | 37
  ≥ TEAE related to study drug | 34
  ≥ 1 NCI Grade 3 or 4 TEAE related to study drug | 22
  ≥ 1 serious TEAE | 28
  ≥ 1 NCI CTC Grade 3 or 4 serious TEAE | 24
  ≥ 1 serious TEAE related to study drug | 14
  TEAE leading to discontinuation of study drug | 8
  TEAE leading to study drug dose reduction | 7
  TEAE leading to study drug dose interruption | 16
  TEAE leading to dose reduction or interruption | 20
  TEAE leading to death | 7

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC∞) of Azacitidine
Description: Area under the plasma concentration-time curve from time zero to infinity (AUC∞) following multiple doses of Azacitidine on Day 7; if possible, the area under the concentration-time curve from time zero to infinity, calculated by the linear trapezoidal rule and extrapolated to infinity was calculated according to the following equation: AUC∞ = AUCt + (Ct/ λz ), where Ct is the last quantifiable concentration. No AUC extrapolation was performed with unreliable λz. If % AUC extrapolated is ≥ 25%, AUC∞ was not reported.
Time Frame: Timeframe: Day 7 pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: The PK population includes all participants with evaluable azacitidine plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
ng*h/mL | 859.1 (23.4)

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUCt) of Azacitidine
Description: Area under the plasma concentration-time curve from time zero to the last quantifiable time point, calculated by the linear trapezoidal rule when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing.
Time Frame: Timeframe: Day 7 pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: The PK population includes all participants with evaluable azacitidine plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
ng*h/mL | 852.8 (23.3)

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Azacitidine
Description: The observed maximum plasma concentration obtained directly from the observed concentration versus time data.
Time Frame: Timeframe: Day 7 pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: The PK population includes all participants with evaluable azacitidine plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
ng/mL | 972.3 (44.0)

14. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Azacitidine
Description: Time to maximum observed plasma concentration obtained directly from the observed concentration versus time data.
Time Frame: Timeframe: Day 7 pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: The PK population includes all participants with evaluable azacitidine plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
hours | 0.29 (27.65)

15. Secondary Outcome: Terminal Phase of Half-life (T1/2) of Azacitidine
Description: The apparent terminal half-life was calculated according to the following equation t½ = 0.693/λz.
Time Frame: Timeframe: Day 7 pre-dose at 0.25, 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: The PK population includes all participants with evaluable azacitidine plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
hours | 1.0 (38.7)

16. Secondary Outcome: Apparent Total Plasma Clearance (CL/F) of Azacitidine
Description: Apparent total plasma clearance (CL/F) of Azacitidine was calculated as Dose/AUC∞
Time Frame: Timeframe: Days 5 and 6 at predose and Day 7 (pre-dose) at 0.25, 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: The PK population includes all participants with evaluable azacitidine plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
L/hr | 149.6 (29.6)

17. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of Azacitidine
Description: Apparent volume of distribution, was calculated according to the equation: Vd/F = (CL/F)/λz
Time Frame: Timeframe: Day 7 pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: The PK population includes all participants with evaluable azacitidine plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Azacitidine
Number analyzed (Participants) | 12
Liters | 205.3 (32.4)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through 28 days after completion of/discontinuation from the study (maximum time on study drug 244 days)
Arm/Group | Azacitidine
Serious Adverse Events (participants affected / at risk) | 28/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine (N=44)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 3
Splenic infarction (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Caecitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 6
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Abdominal infection (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Biliary tract infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Enterobacter infection (Infections and infestations) | 1
Epiglottitis (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 8
Postoperative wound infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 4
Septic shock (Infections and infestations) | 2
Soft tissue infection (Infections and infestations) | 1
Subdiaphragmatic abscess (Infections and infestations) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Acute monocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebellar haemorrhage (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 3
Sciatica (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine (N=44)
Anaemia (Blood and lymphatic system disorders) | 19
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 19
Neutropenia (Blood and lymphatic system disorders) | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 16
Conjunctivitis (Eye disorders) | 4
Dry eye (Eye disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 17
Diarrhoea (Gastrointestinal disorders) | 17
Dyspepsia (Gastrointestinal disorders) | 3
Gingival bleeding (Gastrointestinal disorders) | 8
Haemorrhoids (Gastrointestinal disorders) | 8
Lip ulceration (Gastrointestinal disorders) | 3
Melaena (Gastrointestinal disorders) | 3
Mouth ulceration (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 17
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 17
Asthenia (General disorders) | 6
Fatigue (General disorders) | 9
Feeling cold (General disorders) | 3
Injection site pain (General disorders) | 5
Malaise (General disorders) | 3
Non-cardiac chest pain (General disorders) | 5
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 23
Gingivitis (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Oral candidiasis (Infections and infestations) | 3
Periodontitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 7
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 3
Procedural pain (Injury, poisoning and procedural complications) | 3
Transfusion reaction (Injury, poisoning and procedural complications) | 7
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 3
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 12
Haemochromatosis (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 13
Hyponatraemia (Metabolism and nutrition disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 17
Headache (Nervous system disorders) | 8
Insomnia (Psychiatric disorders) | 9
Haematuria (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10
Ecchymosis (Skin and subcutaneous tissue disorders) | 7
Petechiae (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 9
Rash pruritic (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Multicenter publication must include input from all Investigators involved in the study and Sponsor before its publication; it has priority over subset (single center) publication during 1 year after study completion; Each Investigator has publication rights after multicenter publication is submitted or 1 year after study completion. Sponsor has the right to comment on the publication and ask for a 90-day delay to protect its intellectual property and/or deletion of any confidential information.